CLINICAL TRIAL: NCT04664881
Title: Home Telemonitoring In Patients After Myocardial Infarction, HELP ME Trial
Brief Title: Home Telemonitoring In Patients After Myocardial Infarction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Joerg Herrmann, MD, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20-001646
Record Dates: First submitted 2020-12-07; First posted 2020-12-11 (Actual); Results first posted 2025-05-11 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-04

CONDITIONS: Myocardial Infarction; Heart Attack
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Control (standard treatment) Group (No Intervention): Participants will receive routine cardiac treatment
- SmartHeart Device Group (Experimental): In addition to routine cardiac treatment, participants will wear the SmartHeart device
  Interventions: Device: SmartHeart Device

INTERVENTIONS:
Device: SmartHeart Device — A body-worn device that allows an individual to immediately transmit a 12-lead ECG from anywhere and anytime, using a smartphone application to a physician's office, hospital or monitoring center where designated on-call staff interpret the ECG and make recommendations.
  Arms: SmartHeart Device Group

SUMMARY:
This study is being done to determine if taking an electrocardiogram (ECG) by a portable device (SmartHeart) followed by a phone call will improve patient outcomes by early recognition of abnormalities and decrease emergency room visits and hospital readmissions compared to standard therapy alone.

ELIGIBILITY:
Inclusion Criteria:

* Acute myocardial infarction, both STEMI and non-STEMI.
* Able to use the home ECG telemonitoring.
* Must have smartphone device with home wi-fi/mobile internet which allows for 24/7 ability to transmit ECG.
* Caring family member who will be able to help/perform the ECG in case the patient won't be able to do it.

Exclusion Criteria:

* No ability to use the device at home/unable to comply with the device instructions
* No smartphone device or home wi-fi/mobile internet which prevent 24/7 ability to transmit ECG
* Cannot download the smartheart app
* No support in home environment
* Out of hospital cardiac arrest: secondary to a non-shockable rhythm, unrelated to an acute coronary syndrome, or with any level of neurologic damage.
* Resident of nursing home or acute care facility
* Uninterpretable ECG at discharge - left bundle branch block (LBBB), pacemaker or implantable cardioverter defibrillator (ICD) with pacing dependence.
* Patients who are planned for staged PCI after the index hospitalization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2020-10-14 (Actual); Primary Completion 2024-05-02 (Actual); Study Completion 2024-05-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joerg Herrmann, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Control (Standard Treatment) Group: Participants received routine cardiac treatment
- SmartHeart Device Group: In addition to routine cardiac treatment, participants wore the SmartHeart device
  SmartHeart Device: A body-worn device that allows an individual to immediately transmit a 12-lead ECG from anywhere and anytime, using a smartphone application to a physician's office, hospital or monitoring center where designated on-call staff interpret the ECG and make recommendations.
Period: Overall Study
Arm/Group | Control (Standard Treatment) Group | SmartHeart Device Group
Started | 98 | 97
Completed | 96 | 84
Not Completed | 2 | 13
Not completed — Withdrawal by Subject | 1 | 8
Not completed — Physician Decision | 0 | 5
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control (Standard Treatment) Group | SmartHeart Device Group | Total
Number analyzed (Participants) | 98 | 97 | 195
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.2 (11.0) | 60.9 (10.2) | 61.5 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 34 | 67
  Male | 65 | 63 | 128
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 91 | 89 | 180
  Unknown or Not Reported | 4 | 5 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 1 | 1 | 2
  White | 96 | 90 | 186
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 6 | 6
Region of Enrollment [Number; unit: participants]
  United States | 98 | 97 | 195

OUTCOME MEASURES:

1. Primary Outcome: Emergency Room Visits
Description: Number of emergency room visits over a period of 90 days after an index hospitalization for an acute myocardial infarction
Time Frame: 90 days after hospital discharge
Measure: Number; unit: Emergency Room Visits
Arm/Group | Control (Standard Treatment) Group | SmartHeart Device Group
Number analyzed (Participants) | 98 | 97
Emergency Room Visits | 40 | 33

2. Primary Outcome: Re-hospitalizations
Description: Number of re-hospitalizations over a period of 90 days after an index hospitalization for an acute myocardial infarction
Time Frame: 90 days after hospital discharge
Measure: Number; unit: Re-Hospitalizations
Arm/Group | Control (Standard Treatment) Group | SmartHeart Device Group
Number analyzed (Participants) | 98 | 97
Re-Hospitalizations | 9 | 11

3. Primary Outcome: Mortality Rate
Description: Number of deaths over a period of 90 days after an index hospitalization for an acute myocardial infarction
Time Frame: 90 days after hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Control (Standard Treatment) Group | SmartHeart Device Group
Number analyzed (Participants) | 98 | 97
Participants | 4 | 3
Statistical Analysis 1: Comparison: Control (Standard Treatment) Group vs SmartHeart Device Group; Test type: Superiority; p = 0.71, Chi-squared, Corrected

4. Primary Outcome: Major Adverse Cardiovascular Events
Description: Number of major adverse cardiovascular events including cardiovascular death and hospitalization for myocardial infarction, unstable angina, repeat revascularization, heart failure, stroke, arrhythmias, and cardiac arrest over a period of 90 days after an index hospitalization for an acute myocardial infarction
Time Frame: 90 days after hospital discharge
Population: The study team did not collect stroke data on any of the participants.
Measure: Number; unit: events
Arm/Group | Control (Standard Treatment) Group | SmartHeart Device Group
Number analyzed (Participants) | 98 | 97
events
  Cardiovascular Death | 1 | 2
  Hospitalization for Myocardial infarction | 1 | 4
  Unstable Angia | 0 | 0
  Repeat Revascularization | 0 | 0
  Heart Failure | 0 | 0
  Arrhythmias | 0 | 4
  Cardiac Arrest | 1 | 2
Statistical Analysis 1: Comparison: Control (Standard Treatment) Group vs SmartHeart Device Group; Cardiovascular Death; Test type: Superiority; p = 0.99, Chi-squared, Corrected
Statistical Analysis 2: Comparison: Control (Standard Treatment) Group vs SmartHeart Device Group; Hospitalization for Myocardial Infarction; Test type: Superiority; p = 0.36, Chi-squared, Corrected
Statistical Analysis 3: Comparison: Control (Standard Treatment) Group vs SmartHeart Device Group; Arrhythmias; Test type: Superiority; p = 0.13, Chi-squared, Corrected
Statistical Analysis 4: Comparison: Control (Standard Treatment) Group vs SmartHeart Device Group; Cardiac Arrest; Test type: Superiority; p = 0.99, Chi-squared, Corrected

ADVERSE EVENTS:
Time Frame: Adverse events were collected from patient consent through study completion, approximately 90 days.
Arm/Group | Control (Standard Treatment) Group | SmartHeart Device Group
All-Cause Mortality (participants affected / at risk) | 4/98 | 3/97
Serious Adverse Events (participants affected / at risk) | 3/98 | 6/97
Other Adverse Events (participants affected / at risk) | 24/98 | 22/97
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (Standard Treatment) Group (N=98) | SmartHeart Device Group (N=97)
Hospitalization for Myocardial Infarction (Cardiac disorders) | 2 (2) | 4 (6)
Arrhythmias (Cardiac disorders) | 0 | 4 (4)
Cardiac Arrest (Cardiac disorders) | 1 (1) | 2 (2)
Heart Failure (Cardiac disorders) | 0 | 0
Repeat Revascularization (Cardiac disorders) | 0 | 0
Unstable Angina (Cardiac disorders) | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (Standard Treatment) Group (N=98) | SmartHeart Device Group (N=97)
Non-Cardiac Chest Pain (General disorders) | 0 (0) | 2 (2)
Rapid Heart Rate (Cardiac disorders) | 0 (0) | 1 (1)
Peripheral Edema (General disorders) | 0 (0) | 1 (1)
Chest Pain (Cardiac disorders) | 8 (9) | 10 (10)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 2 (2)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Scalp Laceration (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
General Weakness (General disorders) | 1 (1) | 0 (0)
Neck Pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Angioedema (Immune system disorders) | 0 (0) | 1 (1)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Diverticulitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 2 (2) | 0 (0)
Shoulder Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Numbness and Tingling in Extremity (Nervous system disorders) | 0 (0) | 1 (1)
Pain and Swelling in Hand (General disorders) | 1 (1) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Bleeding (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Elevated Blood Pressure (Surgical and medical procedures) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Gastrointestional Hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Idiopathic Generalized Epilepsy (Nervous system disorders) | 1 (2) | 0 (0)
Fibula Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pelvic Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Swelling over Left Supraorbital Area (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Mechanical Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Malignant Neoplasm of Colon (Gastrointestinal disorders) | 1 (1) | 0 (0)
Allergic Reaction (Immune system disorders) | 1 (1) | 0 (0)
Supraventricular Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Coronary Artery Disease (Cardiac disorders) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-12-27): https://cdn.clinicaltrials.gov/large-docs/81/NCT04664881/Prot_SAP_000.pdf